CLINICAL TRIAL: NCT03632759
Title: Targeting Beta Cell Dysfunction in Longstanding T1D
Brief Title: Targeting Beta Cell Dysfunction With Liraglutide or Golimumab in Longstanding T1D
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carla Greenbaum, MD (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Carla Greenbaum, MD, Director, Diabetes Program, Benaroya Research Institute
Organization: Benaroya Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB18-044
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide; golimumab

STUDY DESIGN:
Intervention Model Description: two independent open label, proof of concept studies
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liraglutide (Experimental): Participants will receive subcutaneous (SC) liraglutide for 8 weeks
  Interventions: Drug: Liraglutide
- Golimumab (Experimental): Participants will receive subcutaneous (SC) golimumab for 8 weeks
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Liraglutide — Participants will receive subcutaneous (SC) liraglutide for 8 weeks
  Other Names: Victoza
  Arms: Liraglutide
Drug: Golimumab — Participants will receive subcutaneous (SC) golimumab for 8 weeks
  Other Names: SIMPONI
  Arms: Golimumab

SUMMARY:
The purpose of this study is to determine whether 8 weeks of Liraglutide or Golimumab can transiently improve beta cell function in patients with longstanding Type 1 diabetes (T1D) who secrete proinsulin and little/no C-peptide.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 3 years from Type 1 diabetes diagnosis
2. Males and females 18-50 years of age, inclusive
3. Peak MMTT stimulated C-peptide <0.017 pmol/mL
4. Proinsulin levels ≥ 2 pM (either fasting or stimulated)
5. Females of child-bearing potential must be willing to use effective birth control for 12 weeks
6. Willing and able to give informed consent for participation
7. HbA1c ≤ 8.5%

Exclusion Criteria:

1. Concurrent use of non-insulin therapies aimed to control hyperglycemia or use within the past 30 days of screening MMTT (V-2).
2. History of severe reaction or anaphylaxis to human, humanized or murine monoclonal antibodies.
3. Diagnosis of liver disease or elevated hepatic enzymes, as defined by ALT or AST> 1.5 x the upper limit of age-determined normal (ULN) .
4. Females who are pregnant or lactating.
5. Receipt of an immune modulating biologic or investigational drug within 3 months or 5 half-lives before enrollment.
6. History of other clinically significant autoimmune disease needing chronic therapy with biologics or steroids with the exception of celiac and stable thyroid disease.
7. Current use of any medication known to significantly influence glucose tolerance (e.g. oral steroids, atypical antipsychotics, diphenylhydantoin, niacin).
8. Any medical or psychological condition that in the opinion of the principal investigator would interfere with the safe completion of the trial.
9. For Study A (liraglutide)

   1. Any history of pancreatitis or elevated amylase or lipase.
   2. Any personal or family history of thyroid C-cell tumors, including medullary thyroid carcinoma (MTC).
   3. Any personal or family history of multiple endocrine neoplasia syndrome type 2.
   4. Hypersensitivity to liraglutide.
   5. Previous treatment with liraglutide.
   6. Known history of clinically significant gastroparesis.
10. For Study B (golimumab)

    1. Any history of recent (within 3 months) serious bacterial, viral, fungal, or other opportunistic infections.
    2. Any history of demyelinating diseases (such as multiple sclerosis), heart failure, or left ventricular dysfunction.
    3. Serologic evidence of current or past HIV, Hepatitis B, or Hepatitis C.
    4. Positive QuantiFERON or PPD TB test, history of tuberculosis, or active TB infection.
    5. Active infection with EBV, defined by real-time PCR.
    6. Active infection with CMV, defined by real-time PCR.
    7. Any of the following hematologic abnormalities at screening:

       * White blood count <3,000/μL or >14,000/μL
       * Lymphocyte count <500/μL
       * Platelet count <140,000 /μL
       * Hemoglobin <8.5 g/dL
       * Neutrophil count <2,000 cells/μL
    8. Receipt of live vaccine (in the 6 weeks before treatment)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals with peak MMTT stimulated C-peptide >0.017 pmol/mL. | 0-to-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Principal Investigator — Benaroya Research Institute
Locations (2):
- United States (2):
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lord SM, Bahnson HT, Greenbaum CJ, Liljenquist DR, Virostko J, Speake C. Testing a new platform to screen disease-modifying therapy in type 1 diabetes. PLoS One. 2023 Dec 14;18(12):e0293268. doi: 10.1371/journal.pone.0293268. eCollection 2023. PMID 38096190